CLINICAL TRIAL: NCT03963518
Title: Immune-checkpoint Inhibitors and Surrogate Endpoints in Cancer Trials
Brief Title: Immune-checkpoint Inhibitors and Surrogate Endpoints in Cancer Trials (SURROGATE-ICI)
Acronym: SURROGATE-ICI
Status: Completed | Type: Observational
Sponsor: Institut Bergonié (Other)
Collaborators: Institut National de la Santé Et de la Recherche Médicale, France (Other Government)
Responsible Party: Sponsor
Other Study IDs: IB2017-SURROGATE-ICI
Record Dates: First submitted 2019-05-23; First posted 2019-05-24 (Actual); Results first posted 2025-09-15 (Actual); Last update posted 2025-10-06 (Actual); Status verified 2025-09

CONDITIONS: Cancer Treated With Immune-checkpoint Inhibitors
Keywords: cancer; trial; immune-checkpoint inhibitors; meta-analysis
MeSH Terms: conditions — Neoplasms | interventions — Nivolumab; Ipilimumab

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Control: nivolumab monotherapy
  Interventions: Drug: nivolumab monotherapy
- Experimental: nivolumab plus ipilimumab
  Interventions: Drug: nivolumab plus ipilimumab

INTERVENTIONS:
Drug: nivolumab monotherapy — nivolumab monotherapy
  Groups: Control
Drug: nivolumab plus ipilimumab — nivolumab plus ipilimumab
  Groups: Experimental

SUMMARY:
Time to next treatment or death (TNT-D) may be a patient-relevant endpoint in patients treated with immune checkpoint inhibitors. This study investigate

ELIGIBILITY:
previously untreated advanced melanoma patients.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: previously untreated advanced melanoma patients included in a recently published clinical trial
Sampling Method: Non-Probability Sample
Enrollment: 631 (Actual)
Dates: Start 2017-01 (Actual); Primary Completion 2020-12 (Actual); Study Completion 2020-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Carine A Bellera, PhD, Principal Investigator — Institut Bergonié
Locations (1):
- Institut Bergonié, Comprehensive Cancer Center, Bordeaux, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Branchoux S, Bellera C, Italiano A, Rustand D, Gaudin AF, Rondeau V. Immune-checkpoint inhibitors and candidate surrogate endpoints for overall survival across tumour types: A systematic literature review. Crit Rev Oncol Hematol. 2019 May;137:35-42. doi: 10.1016/j.critrevonc.2019.02.013. Epub 2019 Mar 1. PMID 31014514
- [Background] Branchoux S, Sofeu CL, Gaudin AF, Kurt M, Moshyk A, Italiano A, Bellera C, Rondeau V. Time to next treatment or death as a candidate surrogate endpoint for overall survival in advanced melanoma patients treated with immune checkpoint inhibitors: an insight from the phase III CheckMate 067 trial. ESMO Open. 2022 Feb;7(1):100340. doi: 10.1016/j.esmoop.2021.100340. Epub 2021 Dec 17. PMID 34929616

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Control | Experimental
Started | 316 | 315
Completed | 316 | 315
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Control | Experimental | Total
Number analyzed (Participants) | 316 | 315 | 631
Age, Continuous [Mean (Full Range); unit: years] | 59 [25 to 90] | 59 [18 to 88] | 59 [18 to 90]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 114 | 113 | 227
  Male | 202 | 202 | 404
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 316 | 315 | 631

OUTCOME MEASURES:

1. Primary Outcome: Correlation Between Time to Next Treatment or Death (TNT-D) and Overall Survival (OS)
Description: Correlation between Time to next treatment or death (TNT-D) and overall survival (OS) in previously untreated advanced melanoma patients.
Time Frame: 4 years after the start of treatment
Measure: Number (95% Confidence Interval); unit: correlation coefficient
Arm/Group | Control | Experimental
Number analyzed (Participants) | 316 | 315
correlation coefficient | 0.63 [0.59 to 0.67] | 0.66 [0.62 to 0.70]

ADVERSE EVENTS:
Time Frame: up to 4 years after the start of treatment Only all-cause mortality was collected for the purpose of this study. Adverse events (serious and non-serious) were not collected for the purpose of this study.
Description: Adverse events (serious and non-serious) were not collected for the purpose of this study
Arm/Group | Control | Experimental
All-Cause Mortality (participants affected / at risk) | 175/316 | 151/315
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-01-05): https://cdn.clinicaltrials.gov/large-docs/18/NCT03963518/Prot_SAP_000.pdf